CLINICAL TRIAL: NCT07043140
Title: Determining the Effectiveness of Mobile Technology-Assisted Self-Management Training for the Prevention of Lymphedema in Breast Cancer Patients
Brief Title: Mobile Self-Management Training for Lymphedema Prevention
Acronym: lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sevim Dolu, Research Asisstant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nursing Faculty
Record Dates: First submitted 2025-06-10; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema Arm
Keywords: Breast Cancer; Mobile Technology; Lymphedema; Self-Management Training
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: This research will be carried out in two phases: methodological research and single-center randomized controlled experimental research. The population of the study will consist of patients diagnosed with breast cancer who have undergone breast surgery at least one (1) month ago at Inonu University Turgut Özal Medical Center Oncology Hospital in Malatya province and who agree to participate in the study. The sample will consist of patients who meet the study criteria at the specified time and place, volunteer to participate in the study, and will be selected by randomized controlled method using a table of numbers in line with the simple random sampling method. The power analysis for the sample size was performed using Gpower version 3.1.9.2 and the minimum number of subjects required in the experimental and control groups was calculated as 50 people in each group (Type I Error = 0.05; Power of Test = 0.80; Effect Value = 0.5; Safety = 0.95). Considering the possible losses that may occ
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): control group
- Experimental group (Experimental): Mobile application
  Interventions: Other: mobile application

INTERVENTIONS:
Other: mobile application — mobile application for lymphedema information and exercise
  Arms: Experimental group

SUMMARY:
Breast cancer is the most common cancer among women in the world and in our country and affects women negatively in many ways. Depending on the treatment, patients experience serious problems. Especially in patients with sentinel lymph node biopsy and axillary lymph node dissection, lymphedema frequently occurs in the postoperative period. Lymphedema can develop at any time after breast cancer surgery and is difficult to treat once it occurs. Lifelong self-management is essential for breast cancer patients to prevent lymphedema and control or delay its progression. In the literature, it has been reported that patients do not have sufficient information about lymphedema, are not aware that they may have lymphedema in the future and do not receive the necessary support. This study aims to determine the effectiveness of mobile technology supported self-management training for the prevention of lymphedema in patients with breast cancer.

The research will be conducted in two stages, methodological and randomized controlled pretest-posttest design. The population of the study will consist of patients diagnosed with breast cancer who have undergone breast surgery at least three months ago at Inonu University Turgut Özal Medical Center Oncology Hospital in Malatya province and who agree to participate in the study. The sample will consist of 147 people in the first stage and 120 people in the second stage, 60 for each group (experimental and control) determined by power analysis. People will be randomly assigned to the experimental and control groups. The research data will be collected using Personal Information Form, Lymphedema Self-Management Support Scale for Breast Cancer Survivors, Breast Cancer Survivorship Self-Efficacy Scale, Rosenberg Self-Esteem Scale. As a result of the research, it will be determined how the mobile application affects the self-management and self-esteem of breast cancer patients. This mobile application developed in line with the results obtained can be recommended to patients with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a disease in which abnormal breast cells grow out of control and form tumors which, if left uncontrolled, spread throughout the body and can even be fatal. Breast cancer is the most common cancer among women in the world and in our country and affects women physically, psychologically and socially. Local (surgical treatment, radiotherapy) and systemic (chemotherapy, hormone therapy, targeted drug therapy, immunotherapy) methods are used in the treatment of breast cancer. It is usually treated surgically, followed by chemotherapy or radiotherapy or a combination of the two. Patients receiving breast cancer treatment experience serious physical, psychological and social problems depending on the treatment. Especially in patients with sentinel lymph node biopsy and axillary lymph node dissection, lymphedema frequently occurs in the postoperative period.

Lymphedema occurs as a result of primary or secondary lymphatic dysfunction. Primary lymphedema is associated with developmental anomalies of the lymphatic system. Secondary lymphedema, on the other hand, is the type that is frequently encountered and usually seen in the upper extremities after breast cancer treatment approaches. Breast cancer-related lymphedema is a pathologic condition in which protein-rich fluid accumulates in soft tissues due to interruption of lymphatic fluid flow and an increase of 2 cm or more in arm circumference . Breast cancer-related lymphedema is a common complication after treatment. Lymphedema may occur in the arm, trunk or preserved breast . The incidence of lymphedema varies according to the treatment administered, lymphedema diagnostic criteria and follow-up period . In the literature, it is reported that the incidence of lymphedema after breast cancer treatment varies between 24.8% and 90.4% . In long-term prospective studies, it was found that the incidence of lymphedema ranged between 42% in five-year follow-up and 15-54% in three-year follow-up. In the early postoperative period after mastectomy, transient arm edema may occur due to local edema in the surgical field, which does not increase the arm circumference by more than 3 cm. The frequency of transient arm edema is not more than 5%. This is not of much clinical importance and does not require treatment. However, lymphedema may develop months or even years after surgery .Breast cancer-related lymphedema may occur immediately after treatment or may occur years later. Lymphedema formation is related with the degree of axillary dissection. The more lymph nodes are removed, the higher the risk of lymphedema. In the literature, it has been reported that breast cancer-related lymphedema is observed at a higher rate in mastectomy compared to breast conserving surgery.

Breast cancer-related lymphedema, a chronic complication, may develop at any time after breast cancer surgery and is difficult to treat once it occurs. The first stage of treatment consists of decongestive treatment methods such as skin care, manual lymph drainage, compression therapy, and exercises. In the second stage, lifelong self-management is essential for breast cancer patients to prevent lymphedema and control or delay its progression . Self-management is a positive and dynamic process in which a person manages his/her own chronic condition, such as lifestyle changes, symptom control, and treatment adherence. It is used to promote physical and mental health and improve quality of life.

In the literature, it has been reported that breast cancer patients at risk of lymphedema do not have sufficient information about lymphedema and are not aware that they may have lymphedema in the future. However, they also reported that they were not adequately informed about lymphedema before or after surgery. Oncology nurses play a key role in identifying patients with breast cancer at risk of lymphedema, providing comprehensive evaluation and early intervention, coordinating appropriate referrals to interdisciplinary team members for lymphedema management, and supporting patient self-management of lymphedema. However, reasons such as inadequate knowledge of nurses about lymphedema, not considering patient education as their role, lack of specialized nurses in this field, and high workload of nurses may negatively affect lymphedema self-management in breast cancer patients.

Considering all these factors, other opportunities should be offered to patients for lymphedema self-management. Especially in recent years, mobile health-based self-management interventions have become popular with the increase in smartphone use. Mobile health-based self-management interventions have been shown to improve self-management behaviors, functional exercise compliance, self-efficacy, disease-related quality of life, and reduce the incidence of lymphedema and anxiety levels in breast cancer patients. Compared to traditional care, it is emphasized that self-management interventions based on mobile health applications may be more useful in terms of eliminating time and space limitations and may facilitate health care by reaching more people.

Based on this literature, this study aims to determine the effectiveness of mobile technology supported self-management training for the prevention of lymphedema in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:Female patients with primary breast cancer

* Patients with unilateral breast cancer
* Those who had breast cancer surgery at least 1 month ago
* Unilateral mastectomy with axillary lymph node dissection (removal of at least 2 lymph nodes)
* 18 years of age or older
* Patients with a body mass index (BMI) ≤ 30 (pretreatment BMI may be a risk factor for lymphedema)
* Those who have a smartphone and know how to use it
* Those without a defined severe mental disorder
* Those who can speak Turkish and have the ability to read, understand and demonstrate awareness of the work
* Those without vision and hearing problems
* Those without communication problems
* Those who volunteered to participate in the study

Exclusion Criteria:

* Metastatic breast cancer or a history of other cancers
* Cancer recurrence detected during the study
* Those diagnosed with lymphodema
* Patients with bilateral lymph node dissection
* Pregnant or breastfeeding patients
* Previously participated in a similar training program
* Those with a medical condition that prevents them from performing the exercises designed to prevent lymphedema
* Patients who refused to participate in the study
* Reluctance to continue with the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women
Enrollment: 120 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Lymphedema Self-Management Support Scale For Breast Cancer Survivors | up to six months
  The Lymphedema Self-Management Support Scale for Breast Cancer Patients was developed by Fu et al. in 2024 to assess and understand the lymphedema self-management support received by breast cancer survivors. The scale consists of 21 items and 4 sub-dimensions. The 5-point Likert-type scale is scored as 0-not at all, 1-slightly, 2-moderately, 3-much, and 4-more. The total score of the scale is between 0 and 84. The higher the score, the higher the degree of support for lymphedema self-management. The total Cronbach's alpha value of the scale is 0.94 and the sub-dimensions are 0.88 for Basic Management Support, 0.95 for Treatment Management Support, 0.73 for Role Management Support and 0.79 for Emotional Management Support.
Rosenberg Self-Esteem Scale | up to six months
  This scale was developed by Rosenberg in 1963 to assess self-esteem and its Turkish validity and reliability study was conducted by Çuhadaroğlu in 1986. Consisting of 63 items, the scale has 12 sub-dimensions and it is stated that the sub-dimensions can be used separately. In this study, the first "10" items of the scale will be used to measure self-esteem for the purpose of the research. Guttman scaling technique is used in scale scoring. Questions 1, 2, 4, 6, 7 of the 4-point Likert-type scale are positive and scored from 3 to 0, while questions 3, 5, 8, 9, 10 are negative and scored from 0 to 3. The total score range is between 0-30, with a score below 15 indicating low self-esteem. In Çuhadaroğlu's validity and reliability study, Cronbach's alpha value was found to be 0.71.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To preserve the originality of the work